CLINICAL TRIAL: NCT04933890
Title: Real-World Evaluation of the Performance of Eko's Heart Murmur Detection Algorithm When Used by Front-line Healthcare Providers on Geriatric Patients
Brief Title: Detection of Heart Conditions Using Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: Eko Devices, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021.5
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Left Ventricular Dysfunction; Heart Failure
MeSH Terms: conditions — Ventricular Dysfunction, Left; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Use of Eko DUO electronic stethoscope — Auscultation of heart sounds using electronic stethoscope

SUMMARY:
The purpose of this study is to evaluate how Eko AI performs in the real world, front-line setting where the availability of sophisticated, expensive diagnostic tools is limited, and where there is a premium on detecting VHD early in its course.

DETAILED DESCRIPTION:
Echocardiography is the state of the art for diagnosing VHD. However, without an effective pre-screening tool, many echocardiograms ("echos") are being ordered unnecessarily. A recent study found that greater than 66% of all echos performed in the United States do not alter clinical management, while an additional 4% may be deemed inappropriate altogether.

Because of this, echos now make up a disproportionately large segment of healthcare expenditure. Each year, 1 in 5 Medicare enrollees receives an echo at a total cost of $1.2 billion, or 11% of total Medicare spending on imaging services. This is compounded by the fact that an estimated 35 million Americans live in medically underserved areas, where patients must travel an average of 56 miles to see a specialist and receive an echo. This does not encourage compliance, and only adds to cost, lost working hours, and inconvenience.

There is therefore a growing, unmet need for better VHD screening tools. Tools that will consistently, reliably, quickly, and cheaply identify VHD when it is early and asymptomatic, when patients can be managed early and appropriately, and when they are at the lowest risk from an intervention. Such a tool will have a positive impact on the cost of care, patient and provider experience, and healthcare outcomes.

The FDA-cleared Eko CORE and Eko DUO electronic stethoscopes offer clinicians a familiar and inexpensive tool that is widely accepted by patients and providers, while at the same time offer sensors and artificial intelligence technology that can improve screening and detection of medical conditions such as VHD. Both the CORE and the DUO feature sound amplification during auscultation - the CORE also offers active noise cancellation - which improves the ability of the clinician to detect nuanced changes in heart sounds.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults who are 18 years and older
* Able and willing to provide informed consent
* Complete a clinical echocardiogram within 7 days before or after study procedures

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Patients who are hospitalized

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a transthoracic echocardiogram will be enrolled. Patients who are over the age of 60 or who are at risk for heart failure (hypertension, murmur, etc.) will be targeted for enrollment. We will also target patients with a referral diagnosis of dyspnea on exertion, orthopnea, lower extremity edema, and possible heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Single-lead ECG based algorithm development | Within two minutes of device use
  Evaluate performance of single-lead ECG based algorithm to identify individuals with reduced ejection fraction.
Single-lead ECG based algorithm Performance | Within two minutes of device use
  To demonstrate that Eko's murmur detection algorithm outperforms front-line healthcare providers in detecting heart murmurs in real-world use. Collecting data in a point-of-care setting will demonstrate how accurately the algorithm detects murmurs in comparison to an unassisted clinical examination. Algorithm output and clinical determination will be confirmed by echocardiographic ground truth, with the results being blinded until the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Parker Jewish Institute of Health Care and Rehabilitation, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No